CLINICAL TRIAL: NCT05107401
Title: Reducing HIV Stigma to Increase HIV Testing Among Adolescents and Young Adults in Kazakhstan Using a Crowdsourcing Approach
Brief Title: Crowdsourcing to Reduce HIV Stigma Among Adolescents and Young Adults in Kazakhstan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Fogarty International Center of the National Institute of Health (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Alissa Davis, Assistant Professor of Social Work, School of Social Work, Columbia University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: AAAT7871; R21TW012017 (NIH)
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Results first posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Stigma, Social; HIV Testing
Keywords: HIV stigma
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive the digital crowdsourced intervention or standard of care (existing HIV informational materials). We will examine effects of the intervention on reducing HIV stigma and increasing HIV testing.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crowdsourced Intervention (Experimental): The digital crowdsourced intervention will be presented to participants in the intervention arm.
  Interventions: Behavioral: Digital Crowdsourced Intervention to Reduce HIV Stigma among Adolescents and Young Adults
- Standard of Care (No Intervention): Standard HIV informational materials currently used by the Kazakhstan Ministry of Health will be presented to participants in the control arm.

INTERVENTIONS:
Behavioral: Digital Crowdsourced Intervention to Reduce HIV Stigma among Adolescents and Young Adults — Adolescents and young adults will participate in a crowdsourcing contest to create digital materials to reduce HIV stigma in order to increase HIV testing. Entries will be judged by a community judging panel and expert judging panel. Winning entries will be selected for the digital intervention and presented to participants in the intervention arm.
  Arms: Crowdsourced Intervention

SUMMARY:
This project will assess whether a digital crowdsourced intervention can reduce HIV stigma and promote HIV self-testing among adolescents and young adults (AYA). NIH has emphasized the need for research on interventions to reduce HIV-associated stigma and its impact on the prevention and treatment of HIV/AIDS, particularly in low and middle income countries (LMICs). The proposed study has the highest public health significance: it uses a community-based participatory approach to engage local AYA to develop a digital crowdsourced HIV stigma reduction and self-testing intervention to reduce HIV stigma and increase HIV testing.

Study Aim 1: To develop a crowdsourced digital HIV stigma reduction and self-testing intervention targeting AYA in Kazakhstan. Using a community-based participatory approach that engages local adolescents and young adults (AYA) and youth organizations, we will launch a national crowdsourcing contest in which AYA will design multimedia content to reduce HIV stigma in order to promote HIV testing among peers.

Study Aim 2: To pilot test this crowdsourced HIV stigma reduction and self-testing intervention in a preliminary efficacy trial. We will assess the intervention's feasibility and acceptability and obtain preliminary estimates of its effects on decreasing HIV stigma (primary outcome) and increasing HIV testing (secondary outcome) among AYA in Kazakhstan who received the intervention compared to individuals who did not. Participants (n=168) will be randomized 1:1 to: 1) receive the winning multimedia crowdsourced HIV stigma reduction content and a link for HIV self-testing, or 2) receive standard Kazakhstan Ministry of Health HIV informational materials and a link for HIV self-testing.

DETAILED DESCRIPTION:
This project will assess whether a digital crowdsourced intervention can reduce HIV stigma and promote HIV self-testing among adolescents and young adults (AYA). Globally AYA are at increased risk for HIV acquisition. In Eastern Europe and Central Asia (EECA), new HIV infections among 15-24 year old AYA are expected to increase 28% by 2030. In Kazakhstan, one in four HIV infections occur among AYA. Despite the growing HIV burden among AYA in Kazakhstan, this population has some of the lowest HIV testing rates in the country, largely due to stigma. Yet few efforts in Kazakhstan address HIV stigma and the role it plays as a barrier to HIV testing. Digital technologies and crowdsourcing campaigns (i.e., engaging groups of AYA online to address public health challenges and share solutions) are scalable, cost-effective tools that can increase HIV testing services and reduce HIV stigma in low and middle income countries (LMICs) and other resource- constrained settings. Crowdsourcing may be particularly successful among AYA, given their high levels of social media use and technological literacy. Complementing the crowdsourcing approach, mailing HIV rapid test kits can enable AYA to avoid the stigma associated with attending the AIDS Center and overcome transportation barriers.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-24
* Report previous sex with another individual
* Reside in Kazakhstan

Exclusion Criteria:

* Not willing to provide consent or not able to understand study procedures

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 216 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alissa Davis, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Global Health Research Center of Central Asia, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with researchers who request access to the data and obtain appropriate IRB approval.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available to outside investigators after the study investigative team has cleaned and analyzed the data and written their proposed papers.
Access Criteria: Have a proposed plan for data analysis Completed human subjects training Obtained Institutional Review Board approval to access and analyze the data

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adolescents and young adults were recruited online via websites and social media advertisements and in-person at youth events in Almaty, Kazakhstan from January to August 2023. Those who were interested in study participation completed an online screening survey.
Groups:
- Crowdsourced Intervention: The digital crowdsourced intervention developed by adolescents and young adults will be presented to participants in the intervention arm.
Period: Overall Study
Arm/Group | Crowdsourced Intervention | Standard of Care
Started | 111 | 105
Completed | 98 | 93
Not Completed | 13 | 12
Not completed — Lost to Follow-up | 13 | 12

BASELINE CHARACTERISTICS:
Groups:
- Crowdsourced Intervention: The digital crowdsourced intervention will be presented to participants in the intervention arm.
  Digital Crowdsourced Intervention to Reduce HIV Stigma among Adolescents and Young Adults: Adolescents and young adults will participate in a crowdsourcing contest to create digital materials to reduce HIV stigma in order to increase HIV testing. Entries will be judged by a community and expert judging panel. Winning entries will be selected for the digital intervention and presented to participants in the intervention arm.
- Total: Total of all reporting groups
Arm/Group | Crowdsourced Intervention | Standard of Care | Total
Number analyzed (Participants) | 111 | 105 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.1 (2.4) | 19.4 (2.4) | 19.7 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 51 | 116
  Male | 46 | 54 | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Kazakh | 58 | 63 | 121
  Ethnicity: Russian | 37 | 28 | 65
  Ethnicity: Other | 16 | 14 | 30
Region of Enrollment [Number; unit: participants]
  Kazakhstan | 111 | 105 | 216
Sexual Orientation [Count of Participants; unit: Participants]
  Heterosexual | 89 | 77 | 166
  Sexual Minority | 22 | 28 | 50

OUTCOME MEASURES:

1. Primary Outcome: Mean Score Change in Total HIV Stigma Scale
Description: The scale/questionnaire is comprised of 17 items on a 5-point Likert scale (score range from 17-85). Higher scores indicate higher levels of stigma. Outcome will be assessed in mean score change from baseline to 3 months follow-up.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Crowdsourced Intervention | Standard of Care
Number analyzed (Participants) | 98 | 93
units on a scale
  Baseline | 47.48 (0.71) | 47.89 (0.74)
  3 month follow-up | 44.60 (0.75) | 47.32 (0.79)
Statistical Analysis 1: Comparison: Crowdsourced Intervention vs Standard of Care; Separate multilevel linear mixed models were calculated for the overall stigma score and then for each of the stigma subscale scores. The multilevel linear mixed models incorporated fixed effects for time (categorical), study arm, and their interaction and included intercept as a random effect. Models were also adjusted for pre-intervention stigma levels, whether the participant had submitted content to the study contest, prior HIV testing, age, sex at birth, and sexual orientation; Test type: Superiority; p = 0.083, Mixed Models Analysis; Mean Difference (Final Values) = -2.30, 95% CI 2-sided [-4.90 to 0.30] — The statistical values presented are the Estimated Value of Mean Difference between study arms from baseline to the three-month follow-up

2. Secondary Outcome: Mean Change in Perceived HIV Test Stigma
Description: This is a subscale of the Total HIV Stigma scale. It contains 2 items, each on a 1-5 point Likert scale, with a range of 5-10. Higher values indicate higher levels of HIV stigma.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Crowdsourced Intervention | Standard of Care
Number analyzed (Participants) | 98 | 93
units on a scale
  Baseline | 5.92 (0.13) | 5.70 (0.14)
  3 months | 5.19 (0.14) | 5.64 (0.14)
Statistical Analysis 1: Comparison: Crowdsourced Intervention vs Standard of Care; Separate multilevel linear mixed models were calculated for the overall stigma score and then for each of the stigma subscale scores. The multilevel linear mixed models incorporated random fixed effects for time (categorical), study arm, and their interaction and included intercept as a random effect. Models were also adjusted for pre-intervention stigma levels, whether the participant had submitted content to the study contest, age, sex at birth, and sexual orientation; Test type: Superiority; p = 0.032, Mixed Models Analysis; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-1.16 to -0.18] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Mean Change in Perceived HIV Healthcare Stigma Subscale
Description: This is a subscale of the Total HIV Stigma Scale. It contains two items, each on a 1-5 point Likert scale, with a range of 5-10. Higher values indicate higher levels of HIV healthcare stigma.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Crowdsourced Intervention | Standard of Care
Number analyzed (Participants) | 98 | 93
units on a scale
  Baseline | 5.80 (0.14) | 5.90 (0.15)
  3 months follow-up | 5.57 (0.15) | 5.89 (0.16)
Statistical Analysis 1: Comparison: Crowdsourced Intervention vs Standard of Care; Separate multilevel linear mixed models were calculated for the overall stigma score and then for each of the stigma subscale scores. The multilevel linear mixed models incorporated random fixed effects for time (categorical), study arm, and their interaction and included intercept as a random effect. Models were also adjusted for pre-intervention stigma levels, whether the participant had submitted content to the study contest, prior HIV testing, age, sex at birth, and sexual orientation; Test type: Superiority; p = 0.48, Mixed Models Analysis; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.72 to 0.29] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Mean Change in Fear & Judgement HIV Stigma Sub-scale
Description: This is a subscale of the Total HIV Stigma Scale. It consists of 5 items, each on a 1-5 point Likert scale, with a range of 5-25. Higher values indicate higher levels of fear & judgement HIV stigma.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Crowdsourced Intervention | Standard of Care
Number analyzed (Participants) | 98 | 93
units on a scale
  Baseline | 11.12 (0.35) | 11.24 (0.36)
  3 months follow-up | 10.56 (0.36) | 11.08 (0.38)
Statistical Analysis 1: Comparison: Crowdsourced Intervention vs Standard of Care; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.48, Mixed Models Analysis; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-1.49 to 0.29] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Mean Change in Perceived Community HIV Stigma Subscale
Description: This is a subscale of the Total HIV Stigma Scale. It consists of 8 items, each on a 1-5 point Likert-scale, with a range of 6-40. Higher values indicate higher levels of perceived community HIV stigma.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Crowdsourced Intervention | Standard of Care
Number analyzed (Participants) | 98 | 93
units on a scale
  Baseline | 24.65 (0.45) | 25.05 (0.47)
  3 month follow-up | 23.28 (0.47) | 24.74 (0.50)
Statistical Analysis 1: Comparison: Crowdsourced Intervention vs Standard of Care; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.37, Mixed Models Analysis; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-2.60 to 0.51] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Uptake of HIV Self-test
Description: The number of participants who ordered an HIV self-test kit after baseline and by the 3-month follow-up. It is a dichotomous outcome (yes/no).
Time Frame: After baseline and by the 3 month follow-up period
Measure: Count of Participants; unit: Participants
Arm/Group | Crowdsourced Intervention | Standard of Care
Number analyzed (Participants) | 98 | 93
Participants | 30 | 18
Statistical Analysis 1: Comparison: Crowdsourced Intervention vs Standard of Care; We used a generalized linear model using a binomial distribution to examine whether the intervention was associated with increased HIV self-testing uptake in the follow-up period. The model was adjusted for history of HIV testing (pre-intervention testing and testing prior to the study), whether the participant had submitted content to the JasSpark contest, and if the participant had a main intimate partner (e.g., girlfriend/boyfriend, spouse); Test type: Superiority; p = 0.099, Regression, Logistic; Risk Ratio (RR) = 1.13, 95% CI 2-sided [0.98 to 1.32] — The statistical values presented are the relative risk between study arms at the three-month follow-up

7. Post Hoc Outcome: Subgroup Analyses By Sex of Mean Change in Total HIV Stigma Scale
Description: The Total HIV Stigma scale consists of 17 items, each on a 1-5 point Likert scale, with a range of 17-85. Higher values indicate higher levels of HIV stigma.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Females - Crowdsourced Intervention; Males - Crowdsourced Intervention: The digital crowdsourced intervention will be presented to participants in the intervention arm.
  Digital Crowdsourced Intervention to Reduce HIV Stigma among Adolescents and Young Adults: Adolescents and young adults will participate in a crowdsourcing contest to create digital materials to reduce HIV stigma in order to increase HIV testing. Entries will be judged by a community and expert judging panel. Winning entries will be selected for the digital intervention and presented to participants in the intervention arm.
- Females - Standard of Care; Males - Standard of Care: Standard HIV informational materials currently used by the Kazakhstan Ministry of Health will be presented to participants in the control arm.
Arm/Group | Females - Crowdsourced Intervention | Females - Standard of Care | Males - Crowdsourced Intervention | Males - Standard of Care
Number analyzed (Participants) | 65 | 51 | 46 | 54
units on a scale
  Baseline | 47.55 (0.91) | 48.24 (1.06) | 47.44 (1.09) | 47.63 (1.02)
  3 months follow-up | 42.39 (0.96) | 48.17 (1.09) | 47.80 (1.16) | 46.41 (1.12)
Statistical Analysis 1: Comparison: Females - Crowdsourced Intervention vs Females - Standard of Care; Sex was marginally significant in the initial multilevel mixed models, therefore, we examined potential moderation effects of sex on stigma changes. Fixed effects corresponding to the two-way interactions involving sex, time, and/or arm, as well as the three-way interaction of sex, time, and arm, were added to the models; Test type: Superiority; p = 0.012, Mixed Models Analysis — To account for multiple comparisons arising from analyses of moderating effects, the false discovery rate (FDR) was controlled using Benjamini-Hochberg procedures in a tiered approach; Mean Difference (Final Values) = -5.09, 95% CI 2-sided [-8.59 to -1.58] — The statistical values presented are the Estimated Value of Mean Difference in females between study arms from baseline to the three-month follow-up
Statistical Analysis 2: Comparison: Males - Crowdsourced Intervention vs Males - Standard of Care; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.56, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Final Values) = 1.58, 95% CI 2-sided [-2.26 to 5.42] — The statistical values presented are the Estimated Value of Mean Difference in males between study arms from baseline to the three-month follow-up

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 3 months, from baseline assessment to the last follow-up assessment.
Arm/Group | Crowdsourced Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/105
Other Adverse Events (participants affected / at risk) | 0/111 | 0/105

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-12-30): https://cdn.clinicaltrials.gov/large-docs/01/NCT05107401/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT05107401/SAP_001.pdf